CLINICAL TRIAL: NCT07127497
Title: Safety and Efficacy Evaluation of Neoadjuvant Chemotherapy Without Radiotherapy Combined With Sintilimab for Locally Advanced Rectal Cancer: Short-term Results of a Single-arm Phase 2 Trial
Brief Title: Clinical Study on the Safety and Relationship of Sintilimab Combined With Chemotherapy in Neoadjuvant Treatment of Locally Advanced Rectal Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PJ 2025-07-31
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-03

CONDITIONS: Pathological Complete Response; Rectal Cancer; Neoadjuvant Chemoimmunotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- the feasibility of neoadjuvant treatment of locally advanced rectal adenocarcinoma with sintilimab c (Experimental): Sintilimab (3 mg/kg, IV, qd for patients with body weight < 60 kg; 200 mg, IV, qd for patients with body weight ≥ 60 kg) combined with XELOX (oxaliplatin 130 mg/m2, IV, qd + capecitabine 1000 mg/m2, bid, d1 - d14, q21d) for 2-4 courses
  Interventions: Biological: Sintilimab combined with XELOX

INTERVENTIONS:
Biological: Sintilimab combined with XELOX — Sintilimab (3 mg/kg, IV, qd for patients with body weight < 60 kg; 200 mg, IV, qd for patients with body weight ≥ 60 kg) combined with XELOX (oxaliplatin 130 mg/m2, IV, qd + capecitabine 1000 mg/m2, bid, d1 - d14, q21d) for 2-4 courses

SUMMARY:
This study is designed as a single-center, phase II exploratory clinical trial to evaluate the pathological response rate and safety of sintilimab (PD-1 inhibitor) combined with XELOX regimen (oxaliplatin + capecitabine) for neoadjuvant treatment of LARC. The study focuses on the pMMR/MSS patient population and attempts to provide a new treatment option for patients who cannot tolerate radiotherapy or need to preserve organ function.

ELIGIBILITY:
Inclusion Criteria:1. Pathologically confirmed rectal adenocarcinoma (non-special type and special type, including mucinous adenocarcinoma, signet ring cell carcinoma, serrated adenocarcinoma, micropapillary carcinoma, medullary carcinoma, cribriform comedo adenocarcinoma); preoperative imaging confirmed that the stage is 1) rectal cancer T3 and (or) N+ resectable rectal cancer patients; 2) for T4 patients, re-evaluation of resectability must be conducted after the completion of neoadjuvant therapy, and radiotherapy may be used in combination depending on the situation. 2. Age ≥ 18 years old, gender is not limited, ECOG score 0-2 points; 3. Physical condition and organ function allow for major abdominal surgery/4. Agree that the researchers use blood, stool and pathological sections for research during the study; 5. Major organ function meets the following requirements (laboratory test values within 7 days before enrollment must meet the following standards) ① Routine blood examination: (no blood transfusion, no use of granulocyte colony stimulating factor, no use of drug correction within 14 days before screening): a) Neutrophil ≥ 1.5×109/L; b) Platelet ≥ 75×109/L; c) Hemoglobin ≥ 90g/L; ② Biochemical examination: (no albumin transfusion within 14 days before screening): a) Serum creatinine ≤ 1.5×upper limit of normal (ULN), or creatinine clearance> 50 mL/min; b) Serum total bilirubin ≤ 1.5×ULN; c) Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN; ③ Coagulation function: a) International normalized ratio (INR) ≤ 2.3 or prothrombin time (PT) exceeds the normal control range ≤ 6 seconds. 6. Patients are recruited regardless of their programmed death ligand 1 (PD-L1) expression level. -

Exclusion Criteria:1) The tumor has distant metastasis or peritoneal metastasis confirmed by laparoscopy; 2) Patients with other severe immunosuppressive diseases or other malignant tumors; 3) Any condition that affects the intestinal absorption of capecitabine; 4) Severe uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases; severe mental illness; severe respiratory diseases; severe liver and kidney dysfunction; history of unstable angina or myocardial infarction within 6 months; history of cerebral infarction or cerebral hemorrhage within 6 months; continuous use of glucocorticoids within 1 month (except local application); 5) The researcher determines that the patient has other complications that endanger the patient's safety or may affect the completion of the study; 6) Currently or previously received other research drugs or any immunotherapy; 7) Suffering from malignant tumors in other parts within five years; 8) The patient is pregnant or lactating;

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
An exploratory, phase II clinical study on the feasibility of neoadjuvant treatment of locally advanced rectal adenocarcinoma with sintilimab combined with chemotherapy | From enrollment to 2-4 courses (about 4-8 weeks) of adjuvant therapy
  Objective response rate refers to the proportion of patients who achieve complete response (CR) and partial response (PR) among the treated patients within a certain period of time.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China